# <u>e</u>verlinQ Endovascular <u>A</u>ccess <u>Systems Enhancements (EASE-2) Study</u>

Study Protocol: CD-0038

Version 01

Date: August 23, 2017

# **Sponsor:**

TVA Medical, Inc. 7000 Bee Cave Rd., Suite 250 Austin, TX, 78746 USA

Phone: (512) 582-2460

NCT Number: 03708562

NCT Number added post-approval per CT.gov requirement

This protocol contains confidential information and is limited in its distribution to Investigational Staff intending to conduct the study and Ethics Committee reviewing this study.

| ABBREVIATIONS | |
|---|---|
| ACT | Activated clotting time |
| ADE | Adverse device effect |
| AE | Adverse event |
| AVF | Arteriovenous fistula |
| AVG | Arteriovenous graft |
| CKD | Chronic kidney disease |
| CMS | Center for Medicare and Medicaid Services |
| CVC | Central venous catheter |
| DBI | Digital brachial index |
| DUS | Duplex ultrasound |
| EC | Ethics Committee |
| eCRF | Electronic case report form |
| endoAVF | Endovascular arteriovenous fistula |
| EQ VAS | EQ visual analogue scale |
| ESRD | End stage renal disease |
| FFBI | Fistula First Breakthrough Initiative |
| HRQOL | Health Related Quality of Life |
| HTN | Hypertension |
| ICF | Informed consent form |
| IFU | Instructions for Use |
| KDOQI | National Kidney Foundation Kidney Disease Outcomes Quality Initiative |
| RF | Radiofrequency |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SVS | Society for Vascular Surgery |
| USADE | Unanticipated serious device effect |
| USRDS | United States Renal Data System |

| DEFINITIONS | |
|---|---|
| Access site - Device | A site of catheters insertion during index procedure. |
| Access site - Cannulation | A vascular site, as a way to reach the blood for hemodialysis. |
| A mais aware | An X-ray procedure that uses contrast agent and a camera (fluoroscopy) to |
| Angiogram | assess and capture flows or blockages in arteries and veins. |
| <b>Bleeding Diathesis</b> | A disorder that involves the tendency to hemorrhage, or bleed. |
| | A term that includes stages such as mild, moderate and severe loss of |
| Chronic Kidney Disease | kidney function based on the patient's level of glomerular filtration rate |
| | (GFR). |
| | Abandonment of the access is defined as an access that can no longer be |
| | used for two needle prescribed dialysis as it may be unable to provide |
| | adequate flows and/or is deemed unsafe for the patient, and the associated |
| | problem cannot be corrected by any intervention, including medical, |
| endoAVF abandonment – | surgical, or radiological interventions or rest. |
| terminal use of endoAVF | Note: switch to peritoneal dialysis, or a kidney transplant is not considered |
| | an abandonment event. Additionally, if an endoAVF was reported to be |
| | matured; however, veins were too deep for cannulation, or if the endoAVF |
| | was not cannulated due to patient preference, these incidences are not |
| | considered abandonment. |
| | The maintenance in the second of AVE (1-5 - 1 - 2 |
| | The re-intervention rate for endoAVF (defined as any intervention required to maintain or re-establish patency) will be calculated at each available |
| endoAVF related | follow-up visit post index procedure. Diagnostic fistulagram and 2nd stage |
| intervention rate | procedures will not be considered an intervention for the purpose of this |
| | study. |
| | · |
| End Stage Renal Disease | Last stage of Chronic Kidney Disease. When the kidneys stop working |
| | well enough to meet the needs of daily life. |
| Hypercoagulable State | Blood clotting disorder. |
| Maturation of endoAVF | Defined as endoAVF that is free of stenosis or thrombosis, with brachial artery flow of at least 500 ml/min and at least 4 mm vein diameter (as |
| Waturation of endoAvF | measured by duplex ultrasound) OR patient was dialyzed using 2 needles. |
| | incasured by duplex diffasound) or patient was diaryzed using 2 needies. |
| | The number of days between the date of AVF creation and the date of |
| Maturation time | endoAVF maturation (based on primary efficacy endpoint definition of |
| | maturation). |
| Dialysis subject | Subject who was receiving hemodialysis at the time of enrollment. |
| Operator | Person who conducts index procedure. |
| Pre-dialysis subject | Subject who was not receiving dialysis at the time of enrollment. |
| Primary patency | The time from endoAVF creation until any intervention designed to |
| 1 i illiar y patency | maintain or reestablish patency, or endoAVF abandonment. |
| Procedure duration | The sum of the venography time, endoAVF creation time, coil and closure |
| | time. |
| Protocol deviation | Deviation from the approved Study Protocol. |
| Stenosis | For the purposes of the study, stenosis is considered flow limiting |
| ~ COMOSIO | complications that led to fistula closure/abandonment. |
| Thrombosis | For the purposes of the study, thrombosis is considered flow limiting blood |
| | clot that led to fistula closure/abandonment. |

| DEFINITIONS | |
|---|---|
| Target fistula site | The anatomical location in the arm where the endoAVF was attempted. |
| Venogram | An X-ray procedure that uses contrast agent and a camera (fluoroscopy) to assess and capture flows or blockages in veins. |

# **Table of Contents**

| 1. | INTRODUCTION | 6 |
|---------|------------------------------------------|----|
| 1.1 | Purpose | 7 |
| 1.2 | Device Description | 7 |
| 2 | RISKS/BENEFITS | 7 |
| 2.2 | Risks | 8 |
| 2.3 | Minimization of Risk | 9 |
| 3 | STUDY METHODOLOGY | 9 |
| 3.2 | Study Objective | 9 |
| 3.3 | Study Endpoints | 9 |
| 3.4 | Investigational Site Selection | 10 |
| 3.5 | Study Population | 10 |
| 3.5.1 | Inclusion Criteria | 10 |
| 3.5.2 | Exclusion Criteria | 11 |
| 4 | STUDY SCREENING AND FOLLOW-UP PROCEDURES | 11 |
| Table 1 | 1: Schedule of Study Procedures | 12 |
| 4.1 | Informed Consent | 12 |
| 4.2 | Screening Evaluation | 12 |
| 4.2.1 | Duplex Ultrasound | 12 |
| 4.2.2 | Angiography/Venography | 13 |
| 4.3 | Index Procedure | 13 |
| 4.4 | Follow-Up Visits | 13 |
| 4.4.1 | Unscheduled Visit | 13 |
| 4.5 | Patient Disposition | 13 |
| 4.6 | Adverse Events | 14 |
| 4.6.1 | Relationship to Device or Procedure | 15 |
| 5 | DATA ANALYSIS | 15 |
| 6 | REGULATORY OBLIGATIONS | 15 |
| 6.1 | Responsibilities of the EC/EC Approval | 15 |
| 6.2 | Sponsor Obligations | 16 |
| 6.2.1 | Investigator's Documents | 16 |
| 6.3 | Investigator Obligations | 16 |
| 6.4 | Records and Reports | 16 |
| 6.4.1 | Investigator's Reports | 17 |
| 6.4.2 | Sponsor's Reports | 18 |
| 6.5 | Site Training | 18 |
| 6.6 | Protocol Deviations | 18 |
| 6.7 | Site Non-Compliance | 18 |
| 6.8 | Device Accountability | 18 |
| 6.9 | Case Report Form Completion | 19 |
| 6.10 | Monitoring Procedures | |
| DEFEI | DENICES | 20 |

#### 1. INTRODUCTION

End Stage Renal Disease (ESRD) currently affects over 2 million people worldwide. It is projected that the worldwide incidence of ESRD will increase dramatically over the next 10 years, due to the increasing incidence of an aging population, diabetes, hypertension, and obesity. Currently, Renal Replacement Therapy for patients with ESRD consists of either hemodialysis or peritoneal dialysis. The rates of implementation of either hemodialysis or peritoneal dialysis vary widely per country. According to the United States Renal Data System (USRDS), in 2006 hemodialysis accounted for around 60% of Renal Replacement Therapy patients in the US, while peritoneal dialysis accounted for 6-7% of patients in the US and the remainder is kidney transplant patients.

Vascular access is a critical component in the care of patients undergoing hemodialysis. The three methods of long term vascular access available to a patient requiring hemodialysis are: an autogenous arteriovenous access or native arteriovenous fistula (AVF), a prosthetic arteriovenous graft (AVG) or a tunneled dialysis catheter.<sup>3</sup> The AVF has been shown to be superior to AVG and superior to catheter access in terms of both mortality and morbidity.<sup>4,5</sup> In fact, the focus of numerous initiatives worldwide has been to increase the implementation of AVF as the preferred method of vascular access in patients requiring hemodialysis. In 1997, the National Kidney Foundation Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines were published to highlight the importance and to promote the increased placement of AVF. These guidelines and subsequent versions have stressed the importance of proactive identification of patients requiring hemodialysis, and have described procedures and quality initiatives to maximize access longevity. In 2006, the updated KDOQI Guidelines recommended that AVF be constructed in at least 65% of prevalent hemodialysis patients. <sup>7</sup> In addition, the AV Fistula First Breakthrough Initiative (FFBI), a coalition lead by the Center for Medicare and Medicaid Services (CMS) has set a formal goal for AVF construction of 65% in prevalent patients by 2009.8 The Society for Vascular Surgery (SVS) has also approved and sponsored initiatives around the development and publication of reporting standards for hemodialysis access and the development of practice guidelines for hemodialysis access.<sup>9</sup>

An AVF is traditionally created during a surgical procedure under general anesthesia. A surgical incision is made in the forearm or upper arm, followed by identification of target arteries and veins for surgical connection. Frequently, prior to the procedure, the vessels are mapped using duplex ultrasound imaging, allowing for pre-operative vessel diameter measurement and vessel selection. Typically, the radial artery or brachial artery and the cephalic vein or basilic veins are selected. The target vessels are carefully dissected and mobilized, and the vein is transected. An arteriotomy is created, and an anastomosis is sewn between the vein and the artery. After completion, the flow is verified using palpation and ultrasound, and the incision is closed. Over the course of the following 1-3 months, the AVF gradually matures, that is, the vein dilates and accepts increased flow sufficient for hemodialysis.

Though there is widespread agreement that the AVF is the preferred method of vascular access, 28-60% of AVFs do not successfully mature and are rendered unusable for hemodialysis. <sup>10,12</sup> This has unintended consequences for patients in immediate need of hemodialysis, since a tunneled dialysis catheter must often be placed. Catheters are associated with higher morbidity, mortality, and costs and are therefore considered a last resort. <sup>11</sup>

To improve on these results, and decrease the invasiveness of the procedure, a new tool and method for creation of an AVF has been developed, called the everlinQ system. The system uses two devices, one inserted into an artery and the other inserted into a closely-positioned vein. The devices contain magnets that bring a pair of electrodes into alignment. Radiofrequency energy is delivered to the electrodes, cutting and/or coagulating the tissue between the electrodes, creating an AVF. The procedure is facilitated using fluoroscopy and ultrasound imaging, to assist in vessel selection and to verify creation of the AVF. Because the vessels are not dissected and not mobilized, leaving the surrounding tissues intact, the vessels do not need to be sewn together with a traditional surgical technique. This proposed method may facilitate the creation of AVF, while reducing the trauma to the patient and also potentially prevent future venous stenosis thought to arise from surgical trauma. In particular, the goal is to reduce the surgical manipulation of the blood vessels, particularly the veins in the arm, which typically exhibit intimal hyperplasia in surgical AVF. Intimal hyperplasia is believed to be a root cause of failure in surgical AVF and AVG, and this technology and method may help improve the patency and maturity of AVF in patients with ESRD.

#### 1.1 Purpose

This clinical pilot study is being conducted to evaluate the everlinQ System when utilized to create an AVF. An initial pilot study conducted under the EASE protocol demonstrated successful creation and high patency rates of an endoAVF in both the proximal radial and ulnar locations utilizing a concomitant vein percutaneous access location to perform the procedure. This study aims to investigate expansion of the percutaneous venous access location to the superficial system which may provide additional procedural benefit.

## 1.2 **Device Description**

The TVA Medical everlinQ System that will be used in this study is an investigational device, and is not cleared by the FDA or any competent authority for sale in the US or elsewhere.

The everlinQ device is a single-use disposable device. The everlinQ catheter system consists of two flexible, magnetic catheters. One (venous) catheter contains an electrode to deliver radiofrequency (RF) energy, and has a cord that is connected for a remote hand switch. The venous catheter and hand switch, along with a standard grounding pad, connect to a standard electrosurgical unit for the delivery of RF energy. The second (arterial) catheter is a flexible magnetic catheter that contains a backstop for the RF electrode of the venous catheter to interface. Once the catheters are properly inserted and aligned, the magnets contained in each catheter attract to one another, approximating the vessels while simultaneously aligning the electrode with the backstop. RF energy is delivered to the electrode whereby the arterio-venous fistula (AVF) is created.

For additional details regarding device or its principal of operation, please refer to the most current Instruction for Use (IFU).

#### 2 RISKS/BENEFITS

#### 2.1 Benefits

The everlinQ System may facilitate a less-invasive and more reproducible AVF procedure. The everlinQ System may allow the physician to cut and coagulate soft tissues for the creation of an AVF while minimizing surgical incisions. Due to the less-invasive nature of the procedure with the

everlinQ System, the AVF may exhibit improved maturation and patency characteristics compared to historical maturation and patency data. In addition, patient recovery time may be decreased, procedural time may be decreased, and anesthesia may be minimized compared to a conventional surgical AVF procedure.

# 2.2 Risks

Many of the potential risks and complications associated with the everlinQ System and procedure are similar to the risks expected for CKD patients undergoing surgically created arteriovenous fistula (AVF) procedures. The potential risks related to the everlinQ System and procedure are similar to surgical AVF creation and may include but not limited to:

- Bruising
- Numbness, tingling and/or coolness in the fistula extremity
- Thrombosis
- Stenosis
- Failure to mature
- Additional procedures
- Venous hypertension
- Aborted procedure
- Swelling, irritation or pain
- Bleeding/ Hemorrhage
- Hematoma
- Wound problem
- Fever
- Steal Syndrome
- Ischemia
- Embolism
- Infection
- Increased risk of congestive heart failure
- Nerve damage
- Vessel damage
- AVF dihesence
- Pseudoaneurysm
- Compartment Syndrome
- Heart problems such as arrhythmias
- Burns
- Problem due to sedation or anesthesia
- Sepsis
- Infiltration injury during fistula cannulation
- Toxic or allergic reaction
- Electrocution
- Death

Most of these potential risks also exist for creation of standard (surgical) AVFs. There may also be other risks related to use of the everlinQ System and procedure that are not listed or that are not known at this time. This study will help characterize the adverse events associated with the everlinQ System.

# 2.3 Minimization of Risk

To minimize the risks, the everlinQ system has undergone pre-clinical and clinical testing under the EASE study. In addition, all Investigators participating in this clinical study will be trained on the everlinQ procedure which will contribute to minimizing risks associated with the use of the device.

#### 3 STUDY METHODOLOGY

#### 3.1 Study Design

This is a prospective, single-center study to evaluate the everlinQ System when used to create an endoAVF in hemodialysis patients. A total of up to 50 subjects will be enrolled and will undergo an endoAVF creation procedure using the everlinQ System. All subjects may be followed for up to 12 months post index procedure based on Investigator's discretion. The duration of the study is expected to be approximately two (2) years.

# 3.2 **Study Objective**

The primary objective of this clinical study is to evaluate the safety and efficacy of using the everlinQ system for the creation of an endovascular AVF (endoAVF) in patients requiring hemodialysis.

#### 3.3 **Study Endpoints**

Study endpoints will be summarized using descriptive statistics. There are no formal hypothesis tests associated with these endpoints.

- **Technical Success:** Intra-procedural verification that the everlinQ device successfully created an endoAVF as determined by an angiogram, the presence of a bruit that is detected with stethoscope, or presence of thrill, or via Duplex Ultrasound.
- **Procedural Success:** Verification that an endoAVF has been created and remains patent 1-7 Days after the index procedure. Patency will be determined by experienced examiner as the presence of a bruit that is detected with stethoscope, or presence of thrill, or via Duplex Ultrasound, or via angiogram.
- **Fistula Maturation**: Defined as endoAVF that is free of stenosis or thrombosis, with brachial artery flow of at least 500 ml/min and at least 4 mm vein diameter (as measured by duplex ultrasound) OR patient was dialyzed using 2 needles.
- **Time to Fistula Maturation:** The number of days between the date of AVF creation and the date of endoAVF maturation (based on primary efficacy endpoint definition of maturation).
- EndoAVF-related Re-intervention Rate: The re-intervention rate for endoAVF (defined as any intervention required to maintain or re-establish patency) will be calculated at each available follow-up visit post index procedure.

- **Primary Patency**: The primary patency rate will be determined via Kaplan-Meier methods and based on the time of endoAVF creation until any intervention designed to maintain or reestablish patency, or endoAVF abandonment.
- Secondary Patency: The secondary patency rate will be determined via Kaplan-Meier methods and based on the time of endoAVF creation until access abandonment. Abandonment due to renal transplant receipt will not be included in this endpoint assessment. Abandonment of the access is defined as an access that can no longer be used for two needle prescribed dialysis as it may be unable to provide adequate flows and/or is deemed unsafe for the patient, and the associated problem cannot be corrected by any intervention, including medical, surgical, or radiological interventions or rest.
- **Safety:** The percentage of patients who experience one or more serious device-related adverse events during the first 3 months following AVF creation.

# • Additional Exploratory Analysis:

- o Rate of serious procedure-related events will be reported
- o Rate of serious device-related events will be reported
- o Rate of device and/or procedure-related infections
- o Arterial and arterialized vein flow rates and diameters will be reported
- o Other analyses may be reported as needed

# 3.4 <u>Investigational Site Selection</u>

Investigational site selected to participate in this clinical study will be dependent on the Investigator at the site having the necessary resources to fulfill the clinical research requirements outlined in the protocol. These resources include adequate patient population, facilities and support staff to perform the clinical evaluation according to all applicable requirements.

# 3.5 Study Population

Candidates for this study are patients being evaluated for placement of an arteriovenous fistula for chronic hemodialysis. Only patients meeting the inclusion and none of the exclusion criteria who signed Informed Consent Form (ICF) will be enrolled in the study.

#### 3.5.1 Inclusion Criteria

- 1. Eligible for a native arteriovenous fistula.
- 2. Adult (age >18 years old).
- 3. Established, non-reversible kidney failure requiring hemodialysis (including pre-dialysis patients).
- 4. Target vein diameter(s) at fistula site  $\geq 2.0$  mm.
- 5. Target artery diameter at fistula site  $\geq 2.0$  mm.
- 6. Procedural access site artery and vein diameter  $\geq 2.0$  mm.
- 7. At least one superficial outflow vein diameter  $\geq 2.5$  mm and in communication with the perforating vein.
- 8. Estimated life expectancy > 1 year.
- 9. Patient is free of clinically significant conditions or illness within 30 days prior to the AV fistula that may compromise the procedure.
- 10. Presence of an antecubital perforating vein diameter  $\geq 2.0$  mm.

#### 3.5.2 Exclusion Criteria

- 1. Known central venous stenosis or central vein narrowing > 50% based on imaging on the same side as the planned AVF creation.
- 2. Upper extremity venous occlusion(s) and/or vessel abnormality(ies) on the same side as the planned AVF creation that precludes endovascular AVF creation by the everlinQ System as deemed by the interventionalists' clinical judgment.
- 3. Prior surgically created access in the planned treatment location.
- 4. Functioning surgical access in the planned treatment arm.
- 5. Pregnant women.
- 6. New York Heart Association (NYHA) class III or IV heart failure.
- 7. Hypercoagulable state.
- 8. Known bleeding diathesis.
- 9. Immunosuppression, defined as use of immunosuppressive medications used to treat an active condition.
- 10. Documented history of drug abuse including intravenous drugs within six months of AVF creation.
- 11. "Planned" concomitant major surgical procedure within 6 months of enrollment or previous major surgery within 30 days of enrollment.
- 12. Currently being treated with another investigational device or drug.
- 13. Known allergy to contrast dye which cannot be adequately pre-medicated.
- 14. Known adverse effects to sedation and/or anesthesia which cannot be adequately premedicated.
- 15. Patients who do not have an ulnar or radial artery.
- 16. Distance between target artery and vein or other anatomical abnormality will not permit catheters to be introduced, navigated to fistula site, or allow magnets to align vessels sufficiently to create the fistula.
- 17. Evidence of calcification in vessels at the fistula site.
- 18. Evidence of active infections on the day of the index procedure.
- 19. Written informed consent not obtained.

## 4 STUDY SCREENING AND FOLLOW-UP PROCEDURES

Patients are required to undergo a thorough screening evaluation prior to the index procedure and return for evaluations according to the study follow-up schedule indicated in Table 1. Study data will be collected on case report forms (CRFs) provided by the Sponsor. Any site's standard of care tests may be done outside of the study (e.g., prior to study participation).

**Table 1: Schedule of Study Procedures** 

| | | | Post Index Procedure | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Screening | Index<br>Procedure | 1-7<br>Days | 30-45<br>Days | 2 Months<br>(Optional) 1 | 3 Months | 6 Months<br>(Optional) <sup>1</sup> | 12 Month<br>(Optional) <sup>1</sup> |
| Compliance<br>window | -60 to 0 days | Day 0 | 1-7<br>days | 30-45<br>days | Anniversary<br>date + 21 days | Anniversary<br>date + 21 days | Anniversary date + 60 days | Anniversary<br>date + 60 days |
| Informed Consent | X | | | | | | | |
| Inclusion/Exclusion | X | | | | | | | |
| History, Physical<br>Exam, Laboratory<br>Evaluation | X | | | | | | | |
| Ultrasound<br>Evaluation | X | X <sup>1</sup> | X | X | X <sup>1</sup> | X | X <sup>1</sup> | X <sup>1</sup> |
| Angiography/<br>Venography | X <sup>1</sup> | X | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> | X <sup>1</sup> |
| Adverse Events | X | X | X | X | X | X | X | X |
| Dialysis Access<br>Data | | | | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> | X <sup>2</sup> |

<sup>&</sup>lt;sup>1</sup> Optional assessment at the discretion of the Primary Investigator

#### 4.1 Informed Consent

Prior to enrollment, all patients will be informed in detail about the nature of the clinical investigation, as well as its risks, potential benefits, and any anticipated discomforts. All patients must provide written informed consent using Ethics Committee (EC) approved informed consent document.

Proper informed consent should be obtained in accordance with local/country guidelines as needed.

## 4.2 **Screening Evaluation**

All patients considered for enrollment must undergo a thorough screening evaluation prior to the scheduled treatment with the everlinQ System. The screening evaluation includes:

- Collection of demographic data;
- A medical history and physical exam;
- A laboratory evaluation (i.e. blood tests); and
- A duplex ultrasound and optional angiography/venography assessment.

There will be a final assessment of the suitability of the patient's study eligibility due to vascular anatomy or other criteria made at the time of the index procedure and thus, there may be some consented subjects who are determined to be ineligible who will not be enrolled in the study.

#### 4.2.1 **Duplex Ultrasound**

All patients are required to undergo duplex ultrasound assessment during screening. DUS needs to be performed to measure the flow rates and inner diameters of the arteries and veins of the target vessels based on the screening documents provided for the study.

<sup>&</sup>lt;sup>2</sup> Will be obtained after dialysis is initiated using endoAVF created by the everlinQ System.

# 4.2.2 Angiography/Venography

Angiographic or venographic assessment of the suitability of the arteries or veins intended for the endoAVF will be performed during the index procedure and may be performed during follow-up at the discretion of the Investigator.

## 4.3 **Index Procedure**

If a patient presents for the index procedure with an active localized infection, or other medical condition that precludes treatment at this time, the procedure should be delayed until the infection or medical condition is treated and resolved.

If the Investigator is not an experienced user of the everlinQ System, a Sponsor's representative will be present as needed for procedures at each site to provide technical guidance to the Investigator.

## 4.4 Follow-Up Visits

See **Table 1** for required and optional follow-up visits.

#### 4.4.1 Unscheduled Visit

In addition to scheduled follow-up visits, the patient should be instructed to contact the Investigator at any time during the follow-up period if he/she has questions or concerns relating to the procedure or the endoAVF. If the patient returns to the clinic for evaluation related to his/her participation in the study, an Unscheduled Visit evaluation should be performed and this data should be recorded on the Follow-Up Visit Case Report Form.

#### 4.5 **Patient Disposition**

The Patient Disposition Case Report Form should be completed whenever a patient exits the study. This includes patients enrolled in the study who:

- complete the study protocol,
- withdraw from the study,
- are lost to follow-up,
- are deceased.
- have other reason(s) for exiting the study.

# 4.6 Adverse Events

For the purpose of this protocol, an AE will be defined as any adverse medical change (i.e., *de novo* or increased severity in a preexisting condition) from the subject's baseline condition that occurs during the course of the clinical study, after starting treatment, whether considered treatment-related or not. All Adverse Events will be classified using the following definitions.

| AE Type | Definition |
|---|---|
| Serious Adverse<br>Event (SAE) | AE that: a) led to death, b) led to serious deterioration in the health of the subject, that either resulted in 1) a life-threatening illness or injury, or 2) a permanent impairment of a body structure or a body function, or 3) in-patient or prolonged hospitalization, or 4) medical or surgical intervention to prevent life-threatening illness or |
| Adverse Device<br>Effect (ADE) | AE related to the use of study device. NOTE: This definition includes adverse events resulting from insufficient or inadequate IFU, deployment, installation, or operation, or any malfunction of the study device. This definition includes any event resulting from use error or from intentional misuse of the study device. |
| Serious ADE<br>(SADE) | ADE that has resulted in any of the consequences characteristic of a SAE |
| Unanticipated SADE (USADE) | USADE which by its nature, incidence, severity or outcome <u>has not</u> been identified in the current version of the study protocol, IFU, or other study documentation. |
| Anticipated<br>SADE (ASADE) | An effect which by its nature, incidence, severity or outcome has been identified in the study documentation. |

To classify the event, you may follow the steps below (please refer to additional local requirements as needed).

| Is this event: | | | | | |
|---|---|---|---|---|---|
| 1. Serious | | Yes | | No | |
| 2. Study device or procedure related | Yes | | No | Yes | No |
| 3. Unanticipated? | Yes | No | | | |
| Event type is → | USADE | ASADE | SAE | ADE | AE (i.e., non-SAE) |

# 4.6.1 Relationship to Device or Procedure

The investigator will also evaluate the relationship of the adverse event to the everlinQ device or procedure according to the following definitions:

**Definite (YES):** The AE follows a reasonable timing from treatment (or attempted

treatment) with the device and the possibilities of factors other than the device or the index procedure, such as underlying disease, concomitant drugs, or concurrent treatment can be excluded. This includes an AE that

occurs during the index (AVF creation) procedure.

**Probable (YES):** The AE follows a reasonable timing from treatment (or attempted

treatment) with the device and the probability of device or procedure involvement cannot be excluded. However, other factors such as

underlying disease, concomitant medications, or concurrent treatment may

be possible.

**Unlikely (NO):** The AE follows an unlikely timing relationship from treatment (or

attempted treatment) or is more likely due to other factors and there is no definitive information suggesting that it was related to the device or

procedure.

**Not Related (NO):** The AE has no timing relationship from treatment (or attempted treatment)

or it can be explained by other factors, including underlying disease,

concomitant medication, or concurrent treatment.

The investigator will also evaluate the relationship to the everlinQ portion of the procedure using the yes/no definitions above. The everlinQ portion of the procedure only includes insertion, deployment and removal of the everlinQ catheters.

#### 5 DATA ANALYSIS

Data analysis will be primarily descriptive in nature. Continuous variables, such as age, height, weight, will be summarized by the mean, standard deviation, median, minimum and maximum values. Nominal variables, such as gender, ethnicity, presence of co-morbid conditions, will be summarized by the number and percentage of subjects within each category defined by the variable. Summary statistics for discrete variables will consist of the number and percent of responses in each category. Other analyses may be performed as needed.

#### 6 REGULATORY OBLIGATIONS

# 6.1 Responsibilities of the EC/EC Approval

The EC has the main responsibility to oversee the welfare of the subjects entered into this study. The EC, by its approval of the informed consent form, also ensures that the potential subjects are aware of the benefits and risk of participation in the study.

Each site must obtain EC approval and any other Regulatory agency's approval as required by local or country guidelines prior to study initiation. A copy of the approval notification and

the approved study specific patient informed consent must also be kept on file at the site and a copy provided to Sponsor prior to the enrollment of patients. If applicable, written EC approval of any subject's information materials or any advertisement must also be attained prior to their use.

# 6.2 **Sponsor Obligations**

The Sponsor must assume responsibilities that are not limited to the following:

- Provide the Investigator with the necessary information (protocol and IFU) and training required to conduct the investigational study.
- Inform study Investigators of all new information.
- Conduct an evaluation of any USADE and report the result of such evaluation to all reviewing ECs and all participating Investigators within 10 working days of first receiving notice of the event.

# **6.2.1** Investigator's Documents

The following documents will be provided to the study Sponsor by the Investigator prior to initiation of the study.

- A signed and dated Study Agreement.
- Current (within one year) curriculum vitae of the Principal Investigator and all Co-Investigators.
- A copy of the approval letter by the EC for the study protocol and the informed consent.

#### 6.3 Investigator Obligations

Upon signing the Study Agreement, the Investigator agrees to assume the following responsibilities, to keep the required records, and to file the required reports in a timely manner.

The Investigator agrees to:

- Conduct the investigation in compliance with the signed agreement, study protocol, and applicable regulations. Changes to the protocol will only be made after approval by the sponsor and the reviewing EC, or when necessary to protect the safety, rights or welfare of a subject.
- Conduct the investigation in compliance with the EC and other applicable Regulatory agencies.
- Personally conduct or supervise the investigation.
- Ensure that all associates, colleagues and employees assisting in the conduct of the study are informed about their obligations.
- Protect the rights, safety and welfare of research subjects. All subjects must be informed that the device is being used for investigational purposes.
- Assure initial and continuing review of the investigation by an EC.

#### 6.4 Records and Reports

All records and reports pertaining to this protocol are subject to inspection by regulatory agencies and must be retained for at least two years after the date on which the investigation is terminated or completed or for two years after the date that the records are no longer required for the purpose of supporting an application to regulatory agencies for commercial approval of the therapy/claims, or per local regulations, whichever is later.

**6.4.1 Investigator's Reports**The investigator is responsible for the preparation and submission of the reports listed below:

| Report | <b>Submitted to</b> | Description |
|---|---|---|
| Unanticipated Serious Adverse Device Events and Serious Adverse Device Effects | Sponsor & EC | The investigator's report on any unanticipated serious adverse device event (USADE) or serious adverse device effect (SADE) must be submitted within 10 working days after the investigator first learns of the event. |
| Withdrawal of EC approval | Sponsor | The investigator must report a withdrawal of reviewing EC approval within 5 working days. |
| Deviations from<br>Study Protocol | Sponsor & EC | Notification must be made within 5 working days of the occurrence of an emergency deviation (made to protect the life or physical well-being of a subject). If the deviation affects the rights, safety, or welfare of the subjects (and is not an emergency), or the scientific soundness of the investigation, prior approval must be obtained from Sponsor, the reviewing EC and applicable Regulatory Authorities (when required). For all other deviations, prior approval must be obtained from Sponsor. All deviations must be documented on a Protocol Deviation Form. |
| Failure to obtain<br>Consent Form | Sponsor & EC | Notification must be made within 5 working days of use of the device. |

#### 6.4.2 Sponsor's Reports

Sponsor is responsible for the preparation and submission of the reports listed below:

| Report | Submitted to | Description |
|---|---|---|
| Unanticipated Serious Adverse Device Effects | EC & Investigators | Sponsor will report on any unanticipated serious adverse device effect evaluation within 10 working days after receiving notice of the effect. |
| Recall and<br>Device<br>Disposition | EC & Investigators | Notification will be made within 30 working days of Sponsor's request that an investigator return, repair or otherwise dispose of any devices. Such notification will state why the request was made. |
| Notification of<br>Termination or<br>Completion | EC & Investigators | Notification will be made within 30 working days of completion or termination of the investigation. |
| Final Report | EC & Investigators | A final report will be submitted within six months after study completion or termination. |
| Emergency<br>Deviations from<br>Study Protocol | EC | Notification will be made within 5 working days after Sponsor learns of an emergency deviation from the Investigational Plan where the deviation was made to protect the life or physical well-being of a subject. |

# 6.5 <u>Site Training</u>

Sponsor representative(s) will be responsible for site personnel training to ensure that all site personnel have a thorough understanding of the protocol, case report forms and associated study requirements.

A Sponsor's representative(s) will meet with the Investigator at each study site prior to the enrollment of patients for the purpose of reviewing and discussing the protocol and supporting documentation to assure total understanding of the requirements involved in performing the clinical evaluation.

# 6.6 **Protocol Deviations**

A Protocol Deviation CRF must be completed for each deviation from the Study Protocol that occurred at the site (e.g., failure to obtain informed consent, enrolling a patient who does not meet inclusion/exclusion criteria, not performing required testing, missed follow-up visits, etc.).

# 6.7 <u>Site Non-Compliance</u>

Repeated serious protocol deviations will be closely monitored. If excessive deviations or a failure to reduce deviations is noted, the Sponsor reserves the right to suspend study enrollment or terminate the site from the study until a sufficient system is in place at the site to reduce further deviations.

## 6.8 **Device Accountability**

A Device Accountability Log (DAL) will be maintained at the study site. Devices allocated for investigational site use will be recorded in the DAL upon delivery to the study site and will be stored in a secured area until use. No devices will be shipped until EC approvals to begin the study are received by the Sponsor. Site personnel will be responsible for tracking the receipt and disposition of all study devices. All unused study devices must be returned to the Sponsor.

The DAL will be updated as each device is used, opened, or returned. The DAL will contain delivery dates of devices to the site, dates used, returned-to-Sponsor dates and the reason for the return, lot numbers of devices delivered to the site, and the patient ID for all used devices.

# 6.9 Case Report Form Completion

Complete and accurate Case Report Forms (CRFs) must be kept for all patients enrolled in the study. All entries in the CRFs should be made with black or blue ink. There must be an entry for every data point in the CRFs. Corrections to the CRFs should be made by striking out the initial entry with a single horizontal line, with placement of the new entry just above the old. All corrections must be initialed and dated by the person making the correction.

All data collected in the study must be supported by source documentation. Source documentation may include, but not necessarily be limited to: patient medical record notes, patient history questionnaires, physical examination forms, duplex ultrasound data, radiology reports, operative summaries or other documentation that is pertinent to the patient's participation in the study. In addition to existing patient records, a copy of the CRF for the study may be used to directly record study data. If the CRF copy is the only documentation of the collection of study data, the copy should be signed and dated by the Investigator and kept in the patient's record as source documentation.

# 6.10 Monitoring Procedures

The Sponsor or a Sponsor representative will monitor the progress of the study as required by GCP. The study data will also be monitored (by utilizing remote risk-based monitoring, if feasible). The Sponsor will request the source documents to be submitted to them in de-identified manner (subject's name and other personal identifiers must be removed and replaced with the study subject identification (ID) number). These source documents may include but not limited to:

- Admission, procedural and discharge reports/notes
- Any documentation relevant to SAE and procedure and device-related AEs

Monitoring will be performed by qualified and appropriately trained monitors onsite and/or remote. They may be Sponsor's employees or Sponsor's representatives.

On-site visits may be performed as needed based upon enrollment, data integrity and site compliance (e.g. repeated and serious non-compliance by the site (significant number of DCFs at the site, etc.). Each remote or on-site monitoring visit will be documented.

#### REFERENCES

- 1. "ESRD 2005 A Worldwide Overview" Wolfgang Meichelboeck, 4<sup>th</sup> International Congress of the Vascular Access Society, Berlin, Germany, 2005. www.vascularaccesssociety.com
- 2. United States Renal Data System (USRDS) 2008 Annual Report.
- 3. Sidway, A.N. et al. Recommended standards for reports dealing with arteriovenous hemodialysis access. J. *Vasc. Surgery* Vol 35(3): 603-610 March 2002.
- 4. Xue, J.L. et al. The association of initial hemodialysis type with mortality outcomes in elderly Medicare ESRD patients. *Am J Kidney Disease* Nov;42(5): 1013-9, 2003.
- 5. Dhingra, R.K. Type of vascular access and mortality in U.S. hemodialysis patients *Kid Int* Vol 60: 1443-1451, 2001.
- 6. National Kidney Foundation. KDOQI guidelines. http://www.kidney.org/professionals/KDOQI/guideline\_upHD\_PD\_VA/index.htm. Accessed: Aug 30, 2009.
- 7. National Kidney Foundation KDOQI 2006 Vascular Access Guidelines. *Am J Kidney Disease* 2006:48(suppl 1):S177-322.
- 8. Fistula First National Vascular Access Improvements Initiative. Available at: <a href="http://www.fistulafirst.org/">http://www.fistulafirst.org/</a>. Accessed August 30, 2009.
- 9. Sidway A.N. et al. The Society for Vascular Surgery: Clinical practice guidelines for surgical placement and maintenance of arteriovenous hemodialysis access. *J Vasc Surgery* Vol 48(5S): 2S-25S, 2008.
- 10. Asif, Roy-Chaudhury, Beathard, G. Early Arteriovenous Fistula Failure: A Logical Perspective of How and Why to Intervene. *Clin J Am Soc Nephrol* 1: 332–339, 2006.
- 11. Schwab, J., Beathard, G. The hemodialysis catheter conundrum: Hate living with them, but can't live without them. *Kidney International* Vol 56:1-17, 1999.
- 12. Dember, L., Beck, G., Allon, M., et al. Effect of Clopidogrel on Early Failure of Arteriovenous Fistulas for Hemodialysis: A Randomized Controlled Trial. JAMA 299(18):2164-2171, 2008.